CLINICAL TRIAL: NCT04893031
Title: Effect of Tocilizumab on Intensive Care Patients With COVID-19 Pneumonia, a Retrospective Cohort Study
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Mehtap Pehlivanlar Küçük, Assistant professor, Colsuntant Intensivist, Karadeniz Technical University
Other Study IDs: 2021/24; 2021-01-24T17_19_44 (Other: Republic of Turkey Ministery of Health)
Record Dates: First submitted 2021-05-10; First posted 2021-05-19 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Tocilizumab; COVID-19; Critical Care; Mortality
Keywords: tocilizumab; COVID-19; Critical Care; Mortality
MeSH Terms: conditions — COVID-19 | interventions — tocilizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tocilizumab treatment group: Symptoms of hypoxia and systemic inflammation (SpO2 <90% on room air with accompanying elevation of any two of the systemic inflammatory markers such as CRP, LDH and Ferritin) and / or acute bilateral infiltrations on chest radiography or rapid progression of existing infiltrations, but who did not need mechanical ventilation at admission and were given tocilizumab treatment.
  Interventions: Drug: Tocilizumab
- Standard treatment group: Patients who did not require mechanical ventilation in intensive care admission and did not receive tocilizumab treatment during any period of hospitalization.

INTERVENTIONS:
Drug: Tocilizumab — 400mg or 800 mg IV tocilizumab treatment according to patient clinical severity
  Groups: Tocilizumab treatment group

SUMMARY:
Although its safety and efficacy in the COVID-19 patient population are still unclear, tocilizumab is one of treatment. Tocilizumab is a U.S. Food and Drug Administration approved IL-6 receptor antagonist widely used to treat CRS secondary to the chimeric antigen receptor T cell. In this study the investigators will evaluate the efficacy of Tocilizumab, an IL-6 antagonist administered in the early period in intensive care patients with COVID-19 pneumonia followed by hypoxic and systemic inflammation is predominant, but who do not support mechanical ventilation.

DETAILED DESCRIPTION:
With this study, the investigators will evaluate the efficacy of Tocilizumab, an IL-6 antagonist administered in the early period in intensive care patients with COVID-19 pneumonia followed by hypoxic and systemic inflammation is predominant, but who do not support mechanical ventilation.

With this study, those with signs of hypoxia and systemic inflammation followed by COVID-19 pneumonia (SpO2 <90% on room air together with the elevation of any two of the systemic inflammatory markers such as CRP, LDH and Ferritin) and / or acute bilateral infiltrates on chest radiograph and tocilizumab the patients who received treatment and those who received standard therapy will be compared.

In the study, cases followed up with COVID-19 pneumonia and respiratory failure between March 2020 and March 2021 will be retrospectively evaluated. Tocilizumab was applied as 400 mg - 800 mg iv (depending on weight). A second dose could be given 12-24 h later if the patient's condition had not improved. Primary end point was determined as intensive care mortality.

ELIGIBILITY:
Inclusion Criteria:

* All patients were admitted to intensive care unit, diagnosed with COVID-19 pneumonia

Exclusion Criteria:

* Patients who require mechanical ventilation in intensive care admission
* Cases who received tocilizumab after being intubated during follow-up even though they were not intubated at admission
* patients for whom tocilizumab is contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were diagnosed with COVID-19 and were admitted to intensive care unit
Sampling Method: Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Rates of intensive care mortality in the groups | 28 Day
  all-cause mortality in the patient groups given and not given tocilizumab in the intensive care unit.

SECONDARY OUTCOMES:
Rates of needed of mechanical ventilation in the groups | 28 Day
  Intubation in tocilizumab or standard therapy group assessed by an event-time analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared with researchers if contact with corresponded.
Supporting Information: Study Protocol, SAP
Time Frame: 1 year